CLINICAL TRIAL: NCT05488834
Title: Nurse-led Pain Management in Adult ICU; A Randomised Stepped-Wedge Hybrid Effectiveness Trial
Brief Title: Nurse-led Pain Management in Adult ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz Medical City (Other Government)
Collaborators: Newcastle University (Other); Qassim University (Other)
Responsible Party: Principal Investigator, Majid Alotni, PhD student, Newcastle University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: KingAbdulazizMC
Record Dates: First submitted 2021-06-14; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Pain Management
Keywords: pain; ICU; critical care; nurses; pain assessment; CPOT
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Intervention Model Description: A hybrid effectiveness-implementation design will be used in this study. This study will use type (III) hybrid effectiveness implementation strategy. The Critical Care Pain Observation Tool (CPOT) is a pain scale tool used to assess pain in critically ill patients who are incapable of reporting pain. CPOT will be implemented in the eight adult ICUs, and at the same time, data will be collected to measure the intervention's effectiveness.
Masking Description: A stepped-wedge cluster randomised trial will be used to roll-out the implementation of CPOT (intervention) in a random sequence across groups. When the study starts, all groups will not be exposed to the intervention (control group). The groups are randomised and switched to the intervention at a predetermined moment. At the beginning of the trial, every two ICUs will be clustered in one group, so four groups will be formed. The study will be conducted over six months. In the first month (month 1), all groups will be in the control period, and then at month 2, the intervention will be implemented to the first group over one month, while the other three groups are in the control arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intensive care units (Other): The unit will be subject to the intervention. Data will be collected from all 8 units in the control phase of this study. Units will then be randomised in blocks to the intervention.
  Interventions: Other: Critical-Care Pain Observation Tool

INTERVENTIONS:
Other: Critical-Care Pain Observation Tool — The Critical Care Pain Observation Tool (CPOT) was created to help assess pain in critically ill patients who were unable to self-report pain.
  The CPOT instrument evaluates facial expression, body movement, muscle tension, and compliance with ventilator or vocalisation to evaluate an individual's pain. The total score ranges from 0 to 8, where 8 is the worst pain. Patients are observed for 60 seconds while resting and during nociceptive procedures such as turning or wound dressings to detect any change in behaviour that could indicate pain. Further, the patient must be observed before and at the peak of analgesia medications administered to evaluate pain treatment effectiveness.
  Other Names: CPOT

SUMMARY:
This project is about implementing a pain scale, the Critical Care Pain Observation Tool (CPOT), in ICU settings at King Abdullah Medical City to evaluate its impact on nurse pain assessment and management.

Pain is considered as a significant problem in ICU and the literature shows that 50% of patients in ICU suffer moderate to severe pain and up to 70% of patients experience undetected pain while in ICU. The CPOT is an evidence-based intervention to assess pain among non-verbal patients in ICU settings. A stepped-Wedge Randomised trial will be used to implement the CPOT in 8 ICU in King Abduullah Medical City. Patient chart audits and a survey of ICU nurses will be conducted post implementation.

DETAILED DESCRIPTION:
This project is about implementing a pain scale, Critical Care Pain Observation Tool (CPOT), in 8 adult ICUs in King Abdullah Medical City to evaluate the impact on nurse pain assessment and management.

The literature shows that pain is perceived to be one of the most concerning issues in ICU and that 50% of patients in the ICU suffer moderate to severe pain. In addition, 70% of patients have undetected pain while admitted to ICU. Evidence-based guidelines suggest that CPOT is the most reliable and efficient pain scale tool for non-verbal patients in ICUs, and it is recommended in countries such as the USA, Canada, Australia and New Zealand. The literature suggests that CPOT has a positive impact on frequency of pain assessment.

A Stepped-Wedge Randomised trial will be used to implement the CPOT and at the same time assess the effectiveness of CPOT on pain assessment frequency and management. Patient charts will be audited, and a survey of nurses will be undertaken post CPOT implementation to assess the CPOT acceptability, appropriateness and feasibility.

ELIGIBILITY:
Patient chart audits

Inclusion Criteria:

* Patient's who are 18 years and above
* Patients must be discharged from ICU

Exclusion criteria:

- Patient's who are on muscle relaxants

Nurses survey

Inclusion criteria

* Working in ICU
* Understand English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 880 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Number of documented pain assessments per 24-hour period | 6 months
  How many times pain is documented and reassessed then charted in the medical file for a non-verbal patient over a 24 hour period.

SECONDARY OUTCOMES:
Level of sedation and analgesia | 6 months
  Measurement of the amount of sedation and analgesics administered to patients. For opioids such as Morphine, the Morphine equivalent units (MME) will be used to standardise the level of analgesia given per day. Other opioids will be equalised to Morphine using this formula: MME/day = Dosage X Doses per day X MME conversion Factor (Sinha et al., 2017).
Length of intubation (LOI) | 6 months
  The LOI is the total time a patient was intubated and invasively ventilated.
ICU stay | 6 months
  The ICU stay is the total time in days that the patient was been admitted to the ICU.
Acceptability | 6 months
  To measure the acceptability of the CPOT intervention, the candidate will apply the post-intervention survey and measure how acceptable the CPOT is to nurses working in the ICUs.
Appropriateness | 6 months
  To measure the perceived fit, compatibility or relevance of the CPOT intervention to nurses working in the ICUs using the post-intervention survey.
Feasibility in nursing practice | 6 months
  To measure how feasible it is to implement the CPOT intervention within the ICUs using the post-intervention survey

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz Medical City, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alotni MA, Sim J, Chu G, Guilhermino M, Barker D, Szwec S, Fernandez R. Impact of implementing the critical-care pain observation tool in the adult intensive care unit: A nonrandomised stepped-wedge trial. Aust Crit Care. 2025 Mar;38(2):101129. doi: 10.1016/j.aucc.2024.09.014. Epub 2024 Nov 2. PMID 39489653